CLINICAL TRIAL: NCT07236125
Title: Investigation of the Relationship Between Dietary Nitrate and Oral Microbiota in Children With Primary Hypertension
Brief Title: Dietary Nitrate and the Oral Microbiome in Children With Primary Hypertension
Status: Not yet recruiting | Type: Observational
Sponsor: Yelda Kasımoğlu (Other)
Collaborators: Istanbul University Scientific Research Projects Coordination Unit- Pending (Unknown)
Responsible Party: Sponsor-Investigator, Yelda Kasımoğlu, Assoc. Prof., Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: 2025/169
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Primary Hypertension
Keywords: primary hypertension; oral microbiome; nitrate-reduction bacteria; salivary nitrite; salivary nitrate; pediatric hypertension; Enterosalivary Nitrate Cycle; Adolescent Hypertension; Salivary Microbiome; Nitrate-Nitrite-Nitric Oxide Pathway; Saliva Biomarkers; Endothelial Dysfunction; Blood Pressure in Adolescents; Non-invasive Biomarkers; Saliva-Based Diagnostics
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Unstimulated whole saliva samples will be collected from all participants using sterile collection tubes. Aliquots of each sample will be stored at -80°C for downstream laboratory analyses. These biospecimens will be used for:
  * Genomic DNA extraction for 16S rRNA gene sequencing to characterize the oral microbiota,
  * Quantification of nitrate-reducing bacterial activity,
  * Measurement of salivary biomarkers, including pH, total protein concentration, and lysozyme activity.
  All retained samples contain DNA and will be used exclusively for research analyses within the scope of this protocol. No leftover samples will be used for commercial purposes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with primary hypertension: This group includes adolescents aged 12-18 years who have been clinically diagnosed with primary hypertension based on repeated office blood pressure measurements according to pediatric hypertension guidelines. Participants will undergo standardized assessments including oral examination, blood pressure measurements, salivary collection, and laboratory analyses. Laboratory procedures include: oral microbiota profiling through 16S rRNA gene sequencing, quantification of nitrate-reducing bacterial activity, measurement of salivary pH, total protein concentration, and lysozyme activity. No therapeutic intervention will be administered. All procedures are observational and aim to characterize microbial and biochemical markers associated with primary hypertension.
  Interventions: Other: No active intervention
- Healthy controls: This group includes healthy adolescents aged 12-18 years with no history of primary or secondary hypertension, chronic systemic disease, or regular medication use affecting cardiovascular or oral microbiome physiology. Participants will undergo standard clinical assessments identical to the hypertension group, including oral examination, salivary collection, and blood pressure measurement. Laboratory procedures will include salivary microbiota analysis (16S rRNA sequencing), assessment of nitrate-reducing bacterial activity, salivary pH, total protein concentration, and lysozyme activity. This cohort serves as the normative comparison group to evaluate microbial and biochemical differences associated with primary hypertension. No intervention will be administered.
  Interventions: Other: No active intervention

INTERVENTIONS:
Other: No active intervention — This is an observational study with no active intervention. No drug, device, behavioral, dietary, surgical, or diagnostic intervention is administered to participants. All study procedures, including oral examination, salivary sampling, pH measurement, biochemical tests, and blood pressure assessment, are non-interventional and part of standard clinical evaluation. The study only aims to observe natural variations in oral microbiota composition, nitrate-reducing activity, and blood pressure without changing participants' medical care.

SUMMARY:
Children and adolescents with primary hypertension (high blood pressure without an underlying secondary cause) are at increased risk of cardiovascular disease in adulthood. Recent research suggests that not only the heart and blood vessels, but also the bacteria living in the mouth may play a role in blood pressure regulation. Certain oral bacteria can convert nitrate from food into nitrite and then into nitric oxide, a substance that helps blood vessels relax. If this nitrate-nitrite-nitric oxide pathway is impaired, blood pressure may rise.

This study aims to investigate the relationship between oral microbiota, salivary nitric oxide reductase activity and blood pressure in children and adolescents with primary hypertension compared with healthy peers. We will recruit participants aged 12-18 years who have a diagnosis of primary hypertension and an age- and sex-matched control group without hypertension.

All participants will undergo a non-invasive oral and dental examination and standardized blood pressure measurements. Saliva samples will be collected to measure pH, flow rate, nitrate and nitrite levels, total protein, lysozyme activity and to analyze the composition of oral bacteria using modern DNA-based techniques. Participants and/or their parents will also complete brief questionnaires about diet and general health.

No medication or dietary supplement will be given as part of the study, and no additional blood samples will be taken beyond routine clinical care. The main risk is minimal discomfort related to oral examination and saliva collection. There is no guaranteed direct benefit for participants; however, the results may help us better understand how oral bacteria and salivary nitric oxide pathways are linked to high blood pressure in young people. This knowledge may support the development of new non-invasive strategies for early detection and prevention of hypertension in the future.

DETAILED DESCRIPTION:
Primary hypertension (PH) in children and adolescents is increasingly recognized as a significant public health concern. Epidemiological data from multiple cohorts, including the Young Finns Study and other long-term follow-ups, demonstrate that elevated systolic blood pressure beginning in adolescence predicts endothelial dysfunction, increased carotid intima-media thickness, and a higher lifetime risk of cardiovascular morbidity. Children with PH frequently show early subclinical changes such as impaired flow-mediated dilation, increased arterial stiffness, heightened sympathetic activity, and altered nitric oxide (NO) bioavailability. Despite these findings, the early biological mechanisms that contribute to PH in youth remain insufficiently characterized, and non-invasive biomarkers for early detection are limited.

Recent advances in pediatric cardiovascular science suggest that the nitrate-nitrite-nitric oxide (NO₃- → NO₂- → NO) enterosalivary pathway may play a previously underappreciated role in blood pressure regulation. This pathway relies heavily on commensal oral bacteria capable of reducing dietary nitrate to nitrite, which is then swallowed and converted to NO systemically. Any disruption in this oral microbial nitrate-reducing capacity, whether due to dysbiosis, impaired oral hygiene, inflammation, dietary differences, or ecological shifts during adolescence may diminish NO bioavailability and subsequently raise blood pressure. Several adult studies have shown that antibacterial mouthwashes, changes in oral microbiota composition, and reduced salivary nitrate-reducing activity lead to measurable increases in systolic and diastolic blood pressure. However, pediatric data remain extremely scarce, with no comprehensive metagenomic investigation of oral microbiota in children with PH published to date.

This study is therefore designed to characterise, in detail, the relationships between (i) salivary microbiota composition, (ii) nitrate/nitrite conversion capacity, (iii) salivary biochemical characteristics, and (iv) blood pressure profiles in adolescents aged 12-18 years diagnosed with primary hypertension. Importantly, the project employs non-invasive sampling methods (stimulated and unstimulated saliva), enabling participation from children who may not tolerate venipuncture or invasive sampling procedures, and providing a practical model for future screening tools.

1. Scientific Rationale and Background 1.1. Pediatric Hypertension

   Primary hypertension in youth was once considered rare but now affects up to 3-5% of adolescents globally. It is strongly associated with obesity, insulin resistance, sympathetic overactivation, endothelial dysfunction, and chronic inflammatory states. Although pharmacological treatment is increasingly used, current pediatric guidelines emphasise early identification and non-pharmacological management strategies.

   1.2. Oral Microbiota and Blood Pressure

   The oral cavity hosts over 700 bacterial species, many of which participate in nitrate metabolism. Key nitrate-reducing genera include Veillonella, Neisseria, Rothia, Actinomyces, and Prevotella. Disturbances in these communities due to diet, oral hygiene, frequent mouthwash use, periodontal inflammation, or underlying systemic disease may reduce the efficiency of nitrate reduction.

   Several human trials in adults have demonstrated that:

   mouthwash-mediated suppression of nitrate-reducing bacteria acutely increases blood pressure,

   dietary nitrate supplementation raises salivary nitrite levels and lowers systolic BP,

   individuals with lower nitrate-reducing capacity have higher resting BP.

   However, children fundamentally differ from adults in oral ecology, immune maturation, hormonal shifts during puberty, diet, and salivary gland physiology. Therefore, adult data cannot be extrapolated to pediatric populations.

   1.3. Nitric Oxide, Vascular Function, and Pediatric Risk

   NO is vital for vascular homeostasis. Reduced NO availability contributes to endothelial dysfunction, impaired vasodilation, increased vascular tone, and early arterial stiffness. Several pediatric studies have demonstrated:

   elevated basal NO metabolites in obese children due to chronic low-grade inflammation,

   disrupted NO pathways in children with early metabolic abnormalities,

   correlations between salivary nitrite levels and systemic metabolic markers.

   Yet, no study has simultaneously examined oral microbiome composition + nitrate reductase activity + pediatric hypertension in a unified framework.
2. Study Objectives and Hypotheses Primary Objective

   To determine whether adolescents with primary hypertension exhibit alterations in oral microbiota composition and reduced salivary nitrate-reducing capacity compared with normotensive controls.

   Secondary Objectives

   To quantify salivary nitrate, nitrite, pH, flow rate, total protein, lysozyme activity and correlate these with blood pressure levels.

   To explore associations between oral microbial diversity (alpha/beta diversity metrics) and hypertension status.

   To identify specific bacterial taxa or functional gene pathways (via metagenomic sequencing) associated with impaired nitrate reduction.

   To evaluate whether salivary microbiome features could serve as non-invasive biomarkers for early vascular risk or masked hypertension.

   To explore relationships between nitrate-related pathways and anthropometric measures, oral health indices, diet, and lifestyle.

   Hypotheses

   Children with PH have distinct oral microbial compositions with lower abundance of nitrate-reducing bacteria.

   Reduced nitrate-reducing capacity is associated with lower salivary nitrite, altered NO metabolism, and higher systolic BP.

   Specific microbial signatures may predict masked hypertension and early vascular dysfunction.
3. Study Design

   This is a observational, cross-sectional, non-interventional clinical study. No therapeutic agents or dietary supplements will be administered. All measurements rely on non-invasive, routine pediatric dental and clinical procedures.

   3.1. Participants

   Two groups will be recruited:

   Primary Hypertension Group (PH Group)

   Diagnosed according to AAP and ESH pediatric hypertension criteria.

   Healthy Control Group

   Age- and sex-matched.

   Normotensive based on standardized clinic measurements.

   3.2. Sample size

   Based on prior microbiome variability estimates and effect sizes in adult nitrate-reduction studies, a minimum of 48 participants is planned (24 PH + 24 control). This number is adequate for exploratory metagenomic and metabolite correlations. Power calculations used α=0.05 and β=0.20 for differences in nitrate reduction capacity.
4. Data Collection Procedures 4.1. Blood Pressure Measurement

   Performed using pediatric cuff-adjusted oscillometric devices validated for clinical use.

   Measurements taken after 5 minutes of rest, in a seated position, using three repeated readings.

   4.2. Clinical Oral Examination

   Conducted by a trained pediatric dentist.

   Assessment includes dental caries, gingival status, and plaque presence.

   4.3. Saliva Collection (Unstimulated)

   Unstimulated saliva for baseline nitrate/nitrite measurements, pH, flow rate, total protein.

   Standardized collection times (morning hours, ≥1 hr after eating, drinking, brushing).

   4.4. Laboratory Measurements

   Biochemical analyses

   Nitrate and nitrite concentrations via standardized kits (colorimetric methods).

   Salivary lysozyme activity (innate immunity marker).

   Total protein via BCA assay.

   pH via pH strips.

   Metagenomic DNA Extraction

   Using a microbiome DNA extraction kit ensuring lysis of both Gram-positive and Gram-negative bacteria.

   Library Preparation for NGS

   Metagenomics library preparation kit

   DNA barcoding kit

   Library quantification and normalization using Illumina-based quantification kits.

   Sequencing

   Performed using Illumina MiSeq 2×300 bp paired-end sequencing.

   Quality control steps include fragment size profiles, chimera removal, and adapter trimming.

   Bioinformatics Pipeline

   FASTQ quality filtering using QIIME2 or similar platforms.

   Taxonomic classification using SILVA/Greengenes/HOMD reference databases.

   Functional analysis via PICRUSt2 or equivalent tools.

   Diversity analyses with Shannon, Simpson, Bray-Curtis metrics.
5. Data Management and Quality Assurance 5.1. Data Validation

   All collected data will undergo range checks and logical consistency checks (e.g., BP ranges, anthropometric plausibility).

   Automated scripts will flag inconsistencies for review.

   5.2. Source Verification

   Clinical data will be reviewed against patient charts by trained clinicians.

   Saliva processing forms will be cross-checked with laboratory data.

   5.3. Laboratory QC

   Use of negative/blank controls during DNA extraction and library preparation.

   Duplicate samples for ~10% of participants to assess technical variability.

   Calibration logs for pipettes, thermocyclers, and sequencing equipment.

   5.4. Data Security

   Data stored on institutional encrypted servers behind firewall protection.

   Only authorized team members will have access.
6. Statistical Analysis Plan 6.1. Primary Analysis

   Compare microbial diversity and nitrate-reducing capacity between PH and control groups using:

   Wilcoxon/Mann-Whitney U tests

   PERMANOVA for beta-diversity

   Differential abundance analysis (ANCOM, DESeq2)

   6.2. Secondary Analyses

   Spearman correlations between salivary biochemical markers and systolic/diastolic BP.

   Multiple linear regression adjusting for BMI, diet, oral hygiene habits.

   Exploratory machine-learning models (random forest) to identify predictive microbial features.

   6.3. Missing Data Plan

   Missing biochemical values handled via multiple imputation or complete case analysis.

   Missing microbiome data due to low DNA yield will be documented, not imputed.
7. Ethical Considerations

   This study involves minimal risk. No blood samples, medications, or interventions will be given. Saliva collection is non-invasive and well tolerated. Consent and assent procedures will be conducted according to institutional and national regulations.

   Ethical approval was obtained from the Istanbul University Faculty of Dentistry Clinical Research Ethics Committee at its meeting dated 14/10/2025 and numbered 206.
8. Potential Impact

The project may reveal novel, non-invasive microbial signatures of early vascular risk in adolescents. Findings could support:

early screening tools for masked or mild hypertension,

dietary nitrate-based preventive strategies,

better understanding of the oral microbiome-vascular axis in youth.

ELIGIBILITY:
Inclusion Criteria:

* Applied to the Istanbul University Faculty of Medicine, Department of Pediatric Nephrology,
* Between the ages of 12 and 18,
* Diagnosed with primary hypertension,
* Clinically excluded from secondary hypertension or heart failure,
* No systemic or chronic disease other than hypertension,
* No periodontal disease, dental infection, or oral mucosal disease,
* Not taking regular antihypertensive or other medications for a chronic disease,
* Not having received antibiotic treatment in the last 3 months,
* Patients who have not used mouthwash in the last 3 months,
* Have no allergies to nitrate-rich foods,
* Both male and female patients will be included.

Exclusion Criteria:

* Younger than 12 years of age or older than 18 years of age
* Clinically diagnosed with secondary hypertension or heart failure
* Have a systemic disease
* Have periodontal disease, dental infection, or oral mucosal disease
* Are taking regular antihypertensive medications or other chronic illnesses
* Have received antibiotic treatment within the last 3 months
* Have used mouthwash within the last 3 months
* Are allergic to nitrate-rich foods will not be included in the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be recruited from children and adolescents aged 12-18 years presenting to the Istanbul University Faculty of Dentistry, Department of Pediatric Dentistry, as well as pediatric patients followed by the Pediatric Nephrology Clinic who have been diagnosed with primary hypertension. The study population includes two groups: (1) adolescents with confirmed primary hypertension, not on antihypertensive medication, and (2) age- and sex-matched healthy controls without systemic disease or blood pressure abnormalities. All participants will be systemically healthy, cooperative, and able to provide saliva samples, undergo oral examinations, and complete questionnaire assessments. Recruitment will be consecutive based on clinic attendance, and all participants and their families will be informed about study procedures before enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Microbiota Composition (16S rRNA Sequencing) | Baseline
  Characterization of bacterial community diversity and relative abundance in unstimulated saliva using 16S rRNA gene sequencing. Analysis will include alpha diversity, beta diversity, and differential taxa abundance between groups, with a focus on nitrate-reducing genera such as Neisseria, Rothia, and Actinomyces.

SECONDARY OUTCOMES:
Salivary Nitrate and Nitrite Levels | Baseline (single visit)
  Quantitative measurement of salivary nitrate-to-nitrite conversion capacity using colorimetric assays. The activity of nitrate-reducing oral bacteria will be assessed by determining nitrite concentrations produced in vitro from standardized nitrate substrate under controlled incubation. Higher nitrite output indicates higher nitrate-reductase activity. Values will be compared between primary hypertension patients and healthy controls.
Salivary pH | Baseline
  Salivary acidity/alkalinity measured using validated pH indicator strips immediately after sample collection. Values will be compared between hypertensive and healthy groups.
Salivary Flow Rate | baseline
  Unstimulated salivary flow rate (mL/min) collected over a timed period (5 minutes). Reduced flow may influence oral microbiota composition and nitrate metabolism.
Salivary Lysozyme Activity | baseline
  Quantitative assessment of innate immune enzyme lysozyme using a commercial colorimetric assay. Alterations in antimicrobial enzyme levels may influence microbial ecology.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Faculty of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li D, Nishi SK, Jovanovski E, Zurbau A, Komishon A, Mejia SB, Khan TA, Sievenpiper JL, Milicic D, Jenkins A, Vuksan V. Repeated administration of inorganic nitrate on blood pressure and arterial stiffness: a systematic review and meta-analysis of randomized controlled trials. J Hypertens. 2020 Nov;38(11):2122-2140. doi: 10.1097/HJH.0000000000002524. PMID 32723980
- [Result] Broxterman RM, La Salle DT, Zhao J, Reese VR, Richardson RS, Trinity JD. Influence of dietary inorganic nitrate on blood pressure and vascular function in hypertension: prospective implications for adjunctive treatment. J Appl Physiol (1985). 2019 Oct 1;127(4):1085-1094. doi: 10.1152/japplphysiol.00371.2019. Epub 2019 Aug 15. PMID 31414959
- [Result] Carey RM, Wright JT Jr, Taler SJ, Whelton PK. Guideline-Driven Management of Hypertension: An Evidence-Based Update. Circ Res. 2021 Apr 2;128(7):827-846. doi: 10.1161/CIRCRESAHA.121.318083. Epub 2021 Apr 1. PMID 33793326